CLINICAL TRIAL: NCT04783233
Title: The Use of Chitosan Succinamide (Chitogel CSK-4) Gel as Packing in Tympanoplasty Surgery
Brief Title: Chitogel CSK-4 Gel as Packing in Tympanoplasty Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Physician left practice.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 1685638
Record Dates: First submitted 2021-01-26; First posted 2021-03-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2022-01

CONDITIONS: Tympanoplasty Surgery
Keywords: Chitogel; Tympanoplasty; Support material
MeSH Terms: interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Packing with Gelfoam: Tympanoplasty surgery with fascia graft (either transcanal or post-auricular) will be preformed. The middle ear and external canal will then be packed with Gelfoam.
  Interventions: Biological: Gelfoam
- Packing with Chitosan succinamide: The surgical intervention and tympanoplasty will be performed as normal. The middle ear and external canal will be packed Chitosan succinamide.
  Interventions: Biological: Chitosan succinamide

INTERVENTIONS:
Biological: Chitosan succinamide — Chitogel will be tested for suitability as a packing material in tympanoplasty surgery.
  Other Names: Chitogel; CSK-4
  Groups: Packing with Chitosan succinamide
Biological: Gelfoam — Gelfoam is the current packing material for tympanoplasty surgery.
  Groups: Packing with Gelfoam

SUMMARY:
Little innovation in the material used for middle ear packing has occurred over the past decade, despite the fact that animal models have shown increased acute inflammation and increased fibrosis in the long term histologically. Although Chitosan Succinamide has shown improved wound healing and hemostasis in the nasal cavity mucosa, it has yet to be used as a support material, hemostatic agent, and healing agent in the middle ear. This study will utilize Chitosan Succinamide as an alternative to purified gelatin foam as a support material in primary tympanoplasty surgery.

DETAILED DESCRIPTION:
A prospective cohort study will be performed. Healthy adults (age > 18) with single tympanic membrane perforations who have been offered and agreed to undergo tympanoplasty surgery with fascia graft (either transcanal or post-auricular) will be recruited. The surgical intervention and procedure of tympanoplasty will be performed as normal, however, the packing material will be randomly chosen using a random number generator. The middle ear and external canal will then be packed with either Chitosan Succinamide or Gelfoam. The patients in both groups will be placed on ciprodex post-operatively for 4 weeks. The patients will be seen post-operatively at 1 week for photo documentation and removal of the lateral aspect of CS/CD or Gelfoam. The patients will be seen at 4 weeks for photo documentation and the remainder of packing removal. At 3 months and 1 year the patients will have photo documentation and an audiogram.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Single tympanic membrane perforation

Exclusion Criteria:

* Chronic recurrent infection or otorrhea
* Previous ear surgery for the study ear
* Shellfish allergy
* Cerebral Spinal Fluid (CSF) leak concern

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for primary tympanoplasty surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
External auditory canal healing | Assess healing of auditory canal starting 1 week up to one year following surgery.
  Physician determines exposed bone and inflammatory response
Tympanic membrane healing | Assess healing of auditory canal starting 1 week up to one year following surgery.
  Physician determines failed tympanic membrane healing and inflammatory response.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Wilkerson, MD, Principal Investigator — Physician of Record
Locations (1):
- Ascension Providence Hospital Novi Campus, Novi, Michigan, United States

REFERENCES:
- [Background] Valentine R, Athanasiadis T, Moratti S, Hanton L, Robinson S, Wormald PJ. The efficacy of a novel chitosan gel on hemostasis and wound healing after endoscopic sinus surgery. Am J Rhinol Allergy. 2010 Jan-Feb;24(1):70-5. doi: 10.2500/ajra.2010.24.3422. PMID 20109331
- [Background] Ngoc Ha T, Valentine R, Moratti S, Robinson S, Hanton L, Wormald PJ. A blinded randomized controlled trial evaluating the efficacy of chitosan gel on ostial stenosis following endoscopic sinus surgery. Int Forum Allergy Rhinol. 2013 Jul;3(7):573-80. doi: 10.1002/alr.21136. Epub 2013 Jan 16. PMID 23322408
- [Background] Dogru S, Haholu A, Gungor A, Kucukodaci Z, Cincik H, Ozdemir T, Sen H. Histologic analysis of the effects of three different support materials within rat middle ear. Otolaryngol Head Neck Surg. 2009 Feb;140(2):177-82. doi: 10.1016/j.otohns.2008.10.023. PMID 19201284